CLINICAL TRIAL: NCT01417364
Title: The Effects of Long Term Cyclic Testosterone Administration on Muscle Function and Bone in Older Men
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to identify any qualifying subjects willing to enroll into this study.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-132
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Aging muscle; Testosterone administration; Bone metabolism
MeSH Terms: conditions — Sarcopenia | interventions — testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Testosterone weekly injections continuously (Active Comparator): Testosterone enanthate 100 mg Intramuscular (IM) weekly injections throughout the study
  Interventions: Drug: Testosterone enanthate
- Cyclic testosterone administration (Experimental): Testosterone injections 100 mg. IM weekly for one month alternating with placebo injections weekly for one month throughout the study
  Interventions: Drug: Testosterone enanthate
- Placebo injections (Placebo Comparator): Placebo injections weekly throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone enanthate — 100 mg. IM weekly throughout study
  Arms: Testosterone weekly injections continuously
Drug: Testosterone enanthate — 100 mg IM weekly for one month alternating with placebo injections for one month throughout the study
  Arms: Cyclic testosterone administration
Drug: Placebo — Injected IM weekly throughout study
  Arms: Placebo injections

SUMMARY:
The general hypothesis is that administration of testosterone to healthy, older men for 52 weeks (1 year) following a cycle of 4 weeks of testosterone administration and 4 weeks without testosterone (i.e., monthly cycled regimen) will provide the same gains in muscle strength, muscle mass, and bone density as standard of care (SOC), continuous administration of testosterone for 52 weeks.

DETAILED DESCRIPTION:
The hypothesis is based on data from our current NIA-funded R01 protocol. The investigators treated older men with weekly intramuscular injections of testosterone enanthate (100 mg) for 4 weeks followed by 4 weeks of placebo injections. This 4-week-on, 4-week-off cycled treatment regimen was repeated for 5 cycles (20 weeks). This group was compared with a group of older men who received SOC weekly intramuscular injections of testosterone enanthate (100 mg) for 20 weeks, and another group who received placebo injections. Our preliminary data showed equal gains over placebo in muscle strength and lean body mass in those who received testosterone for 20 weeks, whether SOC continuous or cycled. Moreover, both groups showed greater bone density and markers of bone formation over placebo. In terms of the anabolic actions of testosterone on skeletal muscle in the older men, the investigators found that continuous and cycled administration of testosterone primarily stimulated muscle protein synthesis for the 20 weeks of the study. Cycled testosterone administration enhanced muscle protein synthesis throughout the full 5 cycles of 20 weeks, with no significant loss in muscle protein synthesis during the off-cycle weeks. Additionally, cycled and continuous testosterone administration reduced serum markers of bone resorption compared with placebo. These exciting findings of the benefits of a cycled testosterone regimen in older men represent a novel therapeutic paradigm over the existing SOC approach of continuous administration. The investigators believe the cycled regimen offers a more safe and efficacious approach to combat sarcopenia and osteoporosis with equal anabolic benefit to muscle and bone with only half the dose of testosterone. Critical to the application of this significant paradigm shift in testosterone administration is to determine whether these effects at 20 weeks can persist for the 52 weeks proposed in this study, which represents a treatment duration applicable to the traditional SOC approach.

Thus, the central hypothesis is that cycled administration of testosterone for 52 weeks in healthy, older men will increase muscle function as determined by muscle strength measurements (Biodex dynamometer), lean body mass (DEXA) and muscle volume (MRI), and bone density (DEXA) similar to SOC continuous testosterone administration. Moreover, the investigators anticipate reduced side effects of testosterone administration in the cycled group since they will receive one half the dose over the 52 weeks. The investigators will test the following specific hypotheses in healthy older adults during 52 weeks of cycled, continuous, or placebo testosterone:

1. Cycled and continuous testosterone will increase muscle strength of upper and lower extremities compared with placebo as determined by Biodex dynamometer assessment.
2. Cycled and continuous testosterone will increase lean body mass and muscle volume compared with placebo as determined by DEXA and MRI.
3. Cycled and continuous testosterone will increase bone density compared with placebo as determined by DEXA. The following specific aims will be tested in a randomized double-blind placebo-controlled trial in healthy, older men (60-75 years) undergoing 52 weeks of cycled, continuous, or placebo testosterone:

1. To determine if cycled and continuous testosterone administration increases muscle strength compared to placebo. 2. To determine if cycled and continuous testosterone administration increases lean body mass and muscle volume compared to placebo. 3. To determine if cycled and continuous testosterone administration increases bone density compared to placebo. Our overall goal is to complete a long-term study to determine whether cycled testosterone achieves the same gains in muscle and bone function in older men as SOC, continuous testosterone administration. If our hypothesis is correct, then the investigators will validate an important paradigm shift in testosterone administration in older men that will help combat the disability of sarcopenia and osteoporosis using half the dose of testosterone of the current SOC approach. This reduction is testosterone dose should lessen the side effects and improve the safety of testosterone administration in healthy older men requiring androgen therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 60-75 years
2. Availability of transportation (i.e., subjects must be able to provide their own transportation to UTMB)
3. Mini Mental State Exam Score (MMSE) > 26

Exclusion Criteria:

1. Exclusionary medications will be an anticoagulant (Coumadin) because of the risk of bleeding during the biopsy procedure and weekly injections and glucocorticoids because of the risk of myopathy.
2. Subjects must be able to successfully complete an exercise stress test using the Bruce protocol because the muscle biopsies in the protocol are stressful and muscle strength measurements will be done. Subjects will be excluded without exercise testing with a history of angina that occurs with exertion or at rest or a myocardial infarction within the last 12 months. Subjects that demonstrate ≥0.1 mV horizontal or downsloping ST segment depression, a drop in systolic blood pressure of ≥10 mm Hg millimeters mercury), and/or frequent or repetitive arrhythmias (defined as ≥10 premature ventricular contractions (PVC)/min, or couplets) during the stress test will be excluded.
3. Subjects with a history of stroke will be excluded.
4. Subjects with LDL cholesterol above 200 mg/dL will be excluded because testosterone administration may elevate LDL cholesterol levels further.
5. Diagnosed prostate cancer or prostatic intraepithelial neoplasia (PIN) or, by the Prostate Cancer Risk Calculator, a >30% risk of having overall prostate cancer or >7% risk of having high grade prostate cancer. This is the current exclusion criteria employed by The National Institute on Aging sponsored Testosterone Trial.
6. Men with serum total testosterone concentrations greater than 500 ng/dL will be excluded.
7. Subjects who engage in high intensity exercise training on a regular basis will be excluded.
8. Any subject who has an established major medical illness such as chronic obstructive pulmonary disease, or untreated sleep apnea will be excluded.
9. A hematocrit greater than 51%.
10. Any subject with a blood pressure on three consecutive measurements taken at one week intervals that has a systolic pressure ≥ 160mm Hg or a diastolic blood pressure ≥ 100mmHg will be excluded. Subjects will be included if they are on two or less blood pressure medications and have a blood pressure below these criteria.
11. Any subject with a history of significant liver disorders or a 3-fold elevation of liver function tests (Alk phos, alanine aminotransferase) (ALT), aspartate aminotransferase (AST).
12. Subjects currently taking anti-bone-resorptive agents such as bisphosphonates, parathyroid hormone, or calcitonin will be excluded from the study.
13. Subjects with uncontrolled endocrine or metabolic disease (e.g. liver disease, renal disease, diabetes).
14. Subjects that are HIV-seropositive or have active hepatitis*.
15. Subjects with a history of recent anabolic or corticosteroids use (within 3 months).
16. Subjects with metal fragments or metal devices contained in their bodies.
17. Any other condition or event considered exclusionary by the PI and covering faculty physician.

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | 1 year
  Muscle strength will be measured using a Biodex 4. All strength measures will be normalized by dividing absolute strength by lean muscle mass.
Lean Body Mass and Muscle Volume | 1 year
  Lean body mass will be determined by DEXA and muscle volume by MRI.
Bone density | 1 year
  Bone density will be determined by DEXA.

SECONDARY OUTCOMES:
Assessment of risk factors | 1 year
  Prostate health Complete Blood Count (CBC)/hypertension Serum estradiol Bone fracture risk.
Assessment of Physical Performance | 1 year
  Subjects will complete a timed 400 Molecular Weight (400MWT) at each study session to assess changes in gait speed as a proxy for physical function. In addition subjects will complete Patient Reported Outcomes Information System (PROMIS®) Short Forms addressing questions related to general health, fatigue, and physical functioning
Assessment of muscle signaling | 1 year
  Testosterone can alter skeletal muscle cell signaling. We will measure changes in key signaling proteins in skeletal muscle tissue. We anticipate that testosterone treatment will increase levels of anabolic signaling proteins and suppress levels of catabolic signaling proteins
Assessment of bone metabolism. | 1 year
  Testosterone can decrease rates of bone turnover (net increase of bone formation). We will measure changes in serum markers of bone formation and bone resorption.
Assessment of Inflammation | 1 year
  Testosterone is protective against inflammation. We will measure concentrations of cytokines in blood and muscle tissue.
Assessment of cardiac stiffness | 1 year
  Cardiac stiffness and relaxation will be assessed using echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Medical Branch, Galveston, Galveston, Texas, United States